CLINICAL TRIAL: NCT03437655
Title: Influence of the Composition of Temporary Restorative Material on the Retention Rate and Sensitivity for Provisional Direct Restorations in Vital Teeth - Clinical Study Randomized
Brief Title: Influence of the Composition of Temporary Restorative Material in Vital Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.358.776
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: MTA; Dental Restoration, Temporary
MeSH Terms: interventions — Eugenol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc oxide and eugenol (Active Comparator): Temporary direct restoration with zinc oxide and eugenol.
  Interventions: Procedure: Carie removal; Procedure: Relative isolation; Procedure: Manipulation of the temporary material based on Zinc Oxide and Eugenol; Procedure: Material insertion on the cavity; Procedure: Finishing the temporary direct restoration
- Mineral trioxide aggregate (Active Comparator): Temporary direct restoration with Mineral trioxide aggregate.
  Interventions: Procedure: Carie removal; Procedure: Relative isolation; Procedure: Manipulation of the temporary material based on Mineral trioxide aggregate; Procedure: Material insertion on the cavity; Procedure: Finishing the temporary direct restoration

INTERVENTIONS:
Procedure: Carie removal — Carie removal with a low speed handpiece
Procedure: Relative isolation — Relative isolation with cotton and gauze.
Procedure: Manipulation of the temporary material based on Zinc Oxide and Eugenol — Manipulation of the temporary material based on Zinc Oxide and Eugenol according to the manufacturer's recommendations
  Arms: Zinc oxide and eugenol
Procedure: Manipulation of the temporary material based on Mineral trioxide aggregate — Manipulation of the temporary material based on Mineral trioxide aggregate according to the manufacturer's recommendations
  Arms: Mineral trioxide aggregate
Procedure: Material insertion on the cavity — Material insertion on the cavity according to the manufacturer's recommendations
Procedure: Finishing the temporary direct restoration — Excess cement removal; Occlusal Adjustment; Finishing and polishing.

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, splithmouth, evaluate the success rate (retation rate and dental sensibility) of temporary direct restorations in vital teeth. The composition of the temporary direct restoration (based on Zinc-Oxide with Eugenol; and mineral trioxide aggregate). Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
The confection of temporary direct restoration is still verry commom in dental clinic routine, either by the time required or by biological requirements.The temporary restorations must have sufficient retention and solubility between the consultation intervals to avoid displacement and infiltration; besides being biocompatible to avoid sensitivity. The aim of this study is through a randomized clinical trial, double blind, splithmouth, evaluate the success rate (retention rate and dental sensibility) of temporary direct restoration on vital teeth. The composition of the temporary material (based on Zinc-Oxide with Eugenol; and based on mineral trioxide aggregate) will be evaluated. Twenty-five participants with at least two vital teeth with the need to confection of direct restoration (each participant) will be selected. The teeth will be randomly divided into 2 different groups according to the temporary material composition (Based on Zinc-Oxide with Eugenol; and based on mineral trioxide aggregate). Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers; both genres; presence of at least two teeth with indication of direct restoration; good oral hygiene.

Exclusion Criteria:

* Dentures or orthodontics; presence of periodontal disease and,or parafunctional habits; systemic disease and, or severe psychological; constant use of analgesic and, or anti-inflammatory or allergic response to dental products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-03-20 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Success rate (retention rate and absence of sensibility) of temporary direct restoration with diferents temporary materials with a 15 days of follow up | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Jabbari YS, Al-Rasheed A, Smith JW, Iacopino AM. An indirect technique for assuring simplicity and marginal integrity of provisional restorations during full mouth rehabilitation. Saudi Dent J. 2013 Jan;25(1):39-42. doi: 10.1016/j.sdentj.2012.10.003. Epub 2012 Nov 10. PMID 23960554
- [Background] Arora SJ, Arora A, Upadhyaya V, Jain S. Comparative evaluation of marginal leakage of provisional crowns cemented with different temporary luting cements: In vitro study. J Indian Prosthodont Soc. 2016 Jan-Mar;16(1):42-8. doi: 10.4103/0972-4052.164911. PMID 27134427
- [Background] Fonseca RB, Martins LR, Quagliatto PS, Soares CJ. Influence of provisional cements on ultimate bond strength of indirect composite restorations to dentin. J Adhes Dent. 2005 Autumn;7(3):225-30. PMID 16240963
- [Background] Hill EE, Lott J. A clinically focused discussion of luting materials. Aust Dent J. 2011 Jun;56 Suppl 1:67-76. doi: 10.1111/j.1834-7819.2010.01297.x. PMID 21564117
- [Background] Koumjian JH, Nimmo A. Evaluation of fracture resistance of resins used for provisional restorations. J Prosthet Dent. 1990 Dec;64(6):654-7. doi: 10.1016/0022-3913(90)90290-s. PMID 2079670
- [Background] Mahn E, Rousson V, Heintze S. Meta-Analysis of the Influence of Bonding Parameters on the Clinical Outcome of Tooth-colored Cervical Restorations. J Adhes Dent. 2015 Aug;17(5):391-403. doi: 10.3290/j.jad.a35008. PMID 26525003
- [Background] Qudeimat MA, Alyahya A, Hasan AA. Mineral trioxide aggregate pulpotomy for permanent molars with clinical signs indicative of irreversible pulpitis: a preliminary study. Int Endod J. 2017 Feb;50(2):126-134. doi: 10.1111/iej.12614. Epub 2016 Feb 22. PMID 26841969
- [Background] von Arx T. [Mineral trioxide aggregate (MTA) a success story in apical surgery]. Swiss Dent J. 2016;126(6):573-95. doi: 10.61872/sdj-2016-06-02. French, German. PMID 27377433
- [Background] Young HM, Smith CT, Morton D. Comparative in vitro evaluation of two provisional restorative materials. J Prosthet Dent. 2001 Feb;85(2):129-32. doi: 10.1067/mpr.2001.112797. PMID 11208201